CLINICAL TRIAL: NCT04799431
Title: A Pilot Study of a Neoantigen-Targeted Vaccine Combined With Anti-PD-1 Antibody for Patients With Stage IV MMR-p Colorectal Cancer and Pancreatic Ductal Adenocarcinoma
Brief Title: Neoantigen-Targeted Vaccine Combined With Anti-PD-1 Antibody for Patients With Stage IV MMR-p Colon and Pancreatic Ductal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never started
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Incyte Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2114; IRB00270405 (Other: Johns Hopkins Medicine Internal Review Board); 5P50CA062924 (NIH)
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Cancer Metastatic; Colorectal Cancer Metastatic
Keywords: Neoantigen Vaccines; Anti-PD-1; Retifanlimab; Cancer Vaccines; Immunotherapy; Colon Cancer; Metastatic colon cancer; Pancreatic Ductal Adenocarcinoma (PDAC); Metastatic pancreatic cancer
MeSH Terms: conditions — Colonic Neoplasms; Pancreatic Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoantigen Vaccine with Poly-ICLC adjuvant and Retifanlimab (Experimental): All participants receive this intervention.
  Interventions: Drug: Neoantigen Vaccine with Poly-ICLC adjuvant; Drug: Retifanlimab

INTERVENTIONS:
Drug: Neoantigen Vaccine with Poly-ICLC adjuvant — Neoantigen Vaccine with Poly-ICLC adjuvant will be administered on days 1, 8, 15 and 22. 2 to 5 subcutaneous injections will be administered in the upper thighs, arms and/or back.
  Drug: 0.3 mg per peptide vaccine + 0.5mg Poly-ICLC
  Other Names: Hiltonol® (Poly-ICLC)
Drug: Retifanlimab — 500 mg will be administered as a 30 minute IV. Infusion (-5 min/+15min) on Day 1 of each 28 day cycle every 4 weeks.
  Other Names: INCMGA00012; MGA012

SUMMARY:
Phase 1 study evaluating feasibility, safety, and immune response to a personalized neoantigen vaccine combined with retifanlimab for MMR-p mCRC and mPDAC patients with measurable disease following first-line FOLFIRINOX/FOLFOXIRI (FFX).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Have histologically or cytologically - proven cancer of the pancreas or colon.
* Have tumor lesions amenable to repeated biopsy, and patient's acceptance to have a tumor biopsy of an accessible lesion at baseline and on treatment if the lesion can be biopsied with acceptable clinical risk (as judged by the investigator).
* Measurable disease as per RECIST 1.1.
* Have sufficient and accessible tissue for NGS and immune-phenotyping.
* Have not received any prior systemic therapy in the metastatic setting for PDA or CRC. Patients who have received adjuvant chemotherapy >12 months prior to the diagnosis of metastatic disease may be eligible.
* ECOG performance status 0.
* Life expectancy of greater than 6 months.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Men must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Is a candidate for definitive surgical resection.
* Is unwilling or unable to undergo standard of care therapy.
* Known history or evidence of brain metastases and/or leptomeningeal spread.
* Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, etc.).
* Receiving active immunosuppressive agents or chronic use of systemic corticosteroids within 14 days of vaccine treatment.
* Has active autoimmune disease that has required systemic treatment in the past 5 years, or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Known history or concurrent interstitial lung disease.
* Has a pulse oximetry < 95% on room air.
* Requires the use of home oxygen.
* Infection with HIV or hepatitis B or C.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has been diagnosed with another cancer or myeloproliferative disorder within the past 5 year.
* Has had surgery within 28 days of dosing of investigational agent, excluding minor procedures (dental work, skin biopsy, etc.), celiac plexus block, and biliary stent placement.
* Has received any non-oncology live vaccine therapy used for prevention of infectious diseases within 28 days of study treatment.
* If at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or other substance abuse (including alcohol) that could potentially interfere with adherence to study procedures or requirements.
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Unwilling or unable to follow the study schedule for any reason.
* Are pregnant or breastfeeding.
* Any radiological or clinical pleural effusions or ascites.
* Any peritoneal involvement by the tumor.
* History of malignant small bowel obstruction.
* On parenteral nutrition.
* Any liver metastasis greater than 3 cm or greater than 5 liver metastases.
* Known or suspected hypersensitivity to Hiltonol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who receive at least one dose of personalized neoantigen vaccine | 9 months
  Percentage of patients that receive at least one dose of personalized neoantigen vaccine in the maintenance setting among the total number of patients who achieved disease response (eligible for vaccine generation).
Number of participants experiencing study drug-related toxicities | 2 years
  Number of participants experiencing study drug-related adverse events Grade 3 or higher as defined by CTCAE v5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 | 2 years
  ORR is defined as the number of patients who are administered at least 1 dose of personalized neoantigen vaccine achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at any time during the study. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Objective Response Rate (ORR) per iRECIST | 2 years
  ORR is defined as the number of patients who are administered at least 1 dose of personalized neoantigen vaccine achieving a complete response (iCR) or partial response (iPR) based on the Response Evaluation Criteria in Solid Tumors (Immune-related RECIST (iRECIST) at any time during the study. iCR = disappearance of all target lesions, iPR is =>30% decrease in sum of diameters of target lesions, progressive disease (iPD) is >20% increase in sum of diameters of target lesions, stable disease (iSD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Disease Control Rate (DCR) | 2 months
  DCR is defined as the number of patients achieving a complete response (CR) or partial response (PR) and stable disease (SD) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at 2 months post first vaccination. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Disease Control Rate (DCR) | 6 months
  DCR is defined as the number of patients achieving a complete response (CR) or partial response (PR) and stable disease (SD) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at 6 months post first vaccination. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Disease Control Rate (DCR) | 12 months
  DCR is defined as the number of patients achieving a complete response (CR) or partial response (PR) and stable disease (SD) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) at 12 months post first vaccination. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Progression-free Survival (PFS) per RECIST 1.1 | 4 years
  PFS is defined as the number of months from the date of first personalized vaccine dose to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Progression-free Survival (PFS) per iRECIST | 4 years
  PFS is defined as the number of months from the date of first personalized vaccine dose to disease progression (progressive disease [iPD] or relapse from complete response [iCR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per iRECIST (iPFS) criteria, iCR = disappearance of all target lesions, Partial Response (iPR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (iPD) is >20% increase in sum of diameters of target lesions, Stable Disease (iSD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Overall Survival (OS) | 4 years
  OS will be measured as the number of months from date of first personalized vaccine dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — SKCCC at the Johns Hopkins Medical Institution

IPD SHARING:
Plan to Share IPD: No